CLINICAL TRIAL: NCT05920239
Title: Assessment of the Involvement of the Inferior Glenohumeral Capsuloligamentous Complex in Adhesive Capsulitis Cases Using Shear Wave Elastography: A Study With Magnetic Resonance Imaging Correlation
Brief Title: Shear Wave Elastography in Adhesive Capsulitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Duzce University (Other)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Research Assistant, Uskudar State Hospital
Other Study IDs: SWE1
Record Dates: First submitted 2023-06-14; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Adhesive Capsulitis
Keywords: Magnetic Resonance Imaging; Shear Wave Elastography
MeSH Terms: conditions — Bursitis | interventions — Magnetic Resonance Imaging; Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Individuals who were not suspected of having adhesive capsulitis based on clinical examination and MRI.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Sonoelastography
- Intervention Group: Patients diagnosed with adhesive capsulitis based on evaluations conducted by clinical specialists, primarily in the fields of physical medicine and rehabilitation, orthopedics and traumatology, and confirmed by two experienced radiologists specializing in musculoskeletal imaging through the evaluation of MRI.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI); Diagnostic Test: Sonoelastography

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — MRI imaging is a diagnostic technique that uses magnetic fields and radio waves to create detailed images of the body's internal structures. It provides high-resolution images of soft tissues, organs, and bones, allowing for the detection and evaluation of various medical conditions.Two experienced radiologists specializing in musculoskeletal imaging will evaluate the images obtained through conventional MRI. Cases demonstrating involvement, characterized by findings such as thickening exceeding 4 mm in the inferior glenohumeral capsuloligamentous complex, signal increase indicating edema on fluid-sensitive sequences, and a reduction in axillary recess volume (greater than 0.53 ml), will be included in the study.
Diagnostic Test: Sonoelastography — Sonoelastography is a medical imaging technique that combines ultrasound imaging with elastography. It is used to assess the mechanical properties and stiffness of tissues in the body.The probe will be carefully positioned perpendicular to the anterior part of the glenohumeral capsuloligamentous complex (IGHCC), ensuring no pressure is applied and preventing anisotropy. It will be specifically oriented in the coronal plane towards the axillary recess. The grayscale examination will reveal irregularly thickened and heterogeneous structures at the axillary recess level in the patient group. On the other hand, in the control group, measurements will be taken from the anterior band of the normal, thin, smooth, and homogeneous structure of the IGHCC.

SUMMARY:
This study aimed to evaluate the contribution of sonoelastography in the diagnosis of adhesive capsulitis in patients with a clinical prediagnosis of adhesive capsulitis (AC) and inferior glenohumeral capsuloligamentous complex (IGHCC) involvement demonstrated by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The study will include a total of 30 patients who will be diagnosed with AC based on clinical evaluation by physicians from various clinical departments, including physical medicine and rehabilitation, and orthopedics. The diagnosis will be confirmed by two experienced radiologists specializing in musculoskeletal imaging. Based on clinical evaluation and MRI findings, a control group of 34 individuals without suspected AC will be included. MRI imaging will be performed using a 3 Tesla MRI scanner. Sonoelastography will be performed using a Siemens Acuson-S2000 ultrasound device with a 9L4 (4-9 MHz) linear probe and the Virtual Touch Quantification (VTQ/ARFI) method. Shear wave elastography will be applied to the IGHCC to obtain the mean shear wave velocity (SWV) values. The contribution of sonoelastography in the diagnosis of adhesive capsulitis in patients with a clinical prediagnosis of adhesive capsulitis (AC) and inferior glenohumeral capsuloligamentous complex (IGHCC) involvement will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Having a preliminary diagnosis of Adhesive Capsulitis in Physical Medicine and Rehabilitation or Orthopedics clinic and the diagnosis confirmed by MRI
* Giving consent to participate

Exclusion Criteria:

* Presence of tumor, arthritis, surgical history, or trauma history in the relevant shoulder joint
* Cervical radiculopathy, a central or peripheral neurological deficit in the upper extremity
* Incomplete sequences or inability to evaluate images due to artifacts in MRI imaging
* Presence of pain and/or limited movement to the extent that it hinders positioning or manipulation for ultrasound examination
* Unwillingness to participate in the study voluntarily

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had a preliminary diagnosis of adhesive capsulitis in Physical Medicine and Rehabilitation or Orthopedics clinic later confirmed by MRI.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the Correlation Between MRI Imaging and Sonoelastography Results | 1 day
  This study aims to compare the measurements of intra-articular glenohumeral capsular thickness (IGHCC) using shear wave elastography in two groups: patients with confirmed adhesive capsulitis based on MRI imaging and patients without adhesive capsulitis on MRI imaging. The correlation between the measured shear wave velocity (SWV) values and the diagnosis of adhesive capsulitis will be examined.By comparing the measurements between and within the groups, the correlation of sonoelastography measurements with MRI imaging in healthy individuals and patients will be investigated using statistical methods. Additionally, the potential impact of sonoelastography on the diagnosis of adhesive capsulitis cases will be examined. This study aims to determine the diagnostic value of sonoelastography in adhesive capsulitis and its potential as a complementary tool to MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan H Soylu, M.D., Principal Investigator — Duzce University
Locations (1):
- Üsküdar State Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data will be shared upon reasonable request by the corresponding author.